CLINICAL TRIAL: NCT05939934
Title: Impact of the Mandibular Advancement Device on Sleep Apnea Syndrome During Discontinuation of Treatment with Continuous Positive Airway Pressure: Randomized Controlled Trial
Brief Title: Impact of the Mandibular Advancement Device on Sleep Apnea During CPAP Withdrawal
Acronym: ORTAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49RC23_0078
Record Dates: First submitted 2023-06-13; First posted 2023-07-11 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Sleep Apnea, Obstructive; Endothelial Dysfunction
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): Patients will be ask not to use any OSAS treatment during the 2 weeks of the study (after the CPAP withdrawal)
- mandibular advancement device (Experimental): Patients will be asked to use mandibular advancement device during the 2 weeks CPAP withdrawal
  Interventions: Device: Mandibular advancement device treatment

INTERVENTIONS:
Device: Mandibular advancement device treatment — a titratable thermoplastic mandibular advancement device will be proposed to patient in the experimental group during the 2 weeks of CPAP withdrawal.
  Arms: mandibular advancement device

SUMMARY:
Obstructive sleep apnea hypopnea syndrome (OSAS) is a frequent disease with neuropsychological and cardiovascular (CV) consequences. Continuous positive pressure (CPAP), the main treatment for OSAHS, is effective on the majority of symptoms but restrictive, which can promote non-compliance. Treatment interruptions are often observed in connection with intercurrent events such as nasal obstructions or even when patients are on the move. However, randomized trials have shown that stopping treatment, even for a short time, leads to a recurrence of symptoms and significant CV disturbances (increase in blood pressure, endothelial dysfunction, cardiac repolarization disorders). It seems important to consider strategies that promote therapeutic continuity. The mandibular advancement device (MAD) is an interesting tool in this regard. MAD is as effective as CPAP on symptoms and CV data. The investigators want to assess its effectiveness as a complementary treatment during treatment discontinuation on the main consequences of OSAHS.

DETAILED DESCRIPTION:
Patients are recruited during sleep consultations in the Angers University Hospital pneumology department among patients followed for severe OSAHS and treated with CPAP. All of the scheduled examinations are carried out in the sleep laboratory of the CHU d'Angers.

Patients meeting the inclusion criteria and not having any non-inclusion criteria are randomized to the "MAD" group or to the "control" group. For patients in the "MAD" group, an appointment with a stomatologist is organized to make and adjust a thermo-molded type MAD.

An initial assessment is carried out for all patients during a day hospitalization specific to the study (study of endothelial function, blood pressure, Osler test, ECG, venous and urinary sampling, and completion of the study questionnaires).

Patients are then asked to stop CPAP treatment for two weeks. Patients in the OAM group use OAM during this period. Patients in the control group do not receive any specific treatment for their OSAHS during this period.

After 2 weeks of stopping CPAP, a second assessment, identical to the initial assessment, is carried out for all patients. This assessment is carried out during one night of hospitalization which also allows a PSG to be carried out under OAM or without treatment.

At the end of this assessment, the study is terminated and the patients resume their usual use of CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Patient accepting MAD treatment
* Patient with an apnea-hypopnea index (AHI) greater than 30 events per hour on the initial recording
* Patient with excessive daytime sleepiness during initial treatment (ESE>10)
* Patient treated for more than 12 months by CPAP with average compliance greater than 5 hours per night

Exclusion Criteria:

* Initial severe daytime sleepiness characterized
* OSAS with ≥ 5 central apneas per hour of sleep at baseline recording
* Previously diagnosed severe cardiac and/or respiratory pathology:
* Body mass index ≥ 35 kg/m2
* Known contraindication to OAM treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in subjective sleepiness | before and two weeks after CPAP withdrawal
  Sleepiness assessed using the Epworth Sleepiness Scale

SECONDARY OUTCOMES:
Change in objective sleepiness | before and two weeks after CPAP withdrawal
  Osler test
Change in subjective sleep quality | before and two weeks after CPAP withdrawal
  Pittsburgh sleep quality index
Change in executive function | before and two weeks after CPAP withdrawal
  trail making test
Change in 24 hour blood pressure | before and two weeks after CPAP withdrawal
  24 hours systolic, diastolic and mean blood pressure (Blood pressure holter)
Change in endothelial function | before and two weeks after CPAP withdrawal
  endothelial function (assessed by reactive hyperemia arterial tonometry)
Change in cardiac repolarization | before and two weeks after CPAP withdrawal
  cardiac repolarization (QTc, TpTec intervals calculation on electrocardiographe))
Change in catecholamines levels | before and two weeks after CPAP withdrawal
  urine catecholamines levels
Change in glucose levels | before and two weeks after CPAP withdrawal
  blood glucose levels
Change in Microparticles | before and two weeks after CPAP withdrawal
  blood microparticles levels
Change in oxydative stress | before and two weeks after CPAP withdrawal
  blood 8-isoprostane levels
Change in inflammation | before and two weeks after CPAP withdrawal
  blood CRPus levels

CONTACTS AND LOCATIONS:
Overall Officials: wojciech Trzepizur, MD PHD, Principal Investigator — Angers University Hospital
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: No